CLINICAL TRIAL: NCT06597357
Title: Evaluation of Clinical and Radiographic Outcomes of Meniscal Lesion Treatment Using Collagen Scaffolds (CMI)
Acronym: SUPER CMI
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: SUPER CMI
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Meniscal Degeneration; Osteoarthritis of Knee; Meniscus Injury
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroscopy; Adenosine Monophosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Arthroscopy & saline irrigation alone — the meniscus scaffold is aimed at replacing partial meniscus defect with a synthetic device.

SUMMARY:
Meniscal lesions represent the most frequently encountered joint pathology in the adult population and can cause pain symptoms, mechanical blockages, and recurrent effusions. The treatment of these lesions has progressively evolved from meniscectomy (removal of the damaged meniscal tissue) to the use of meniscal sutures (where possible) to preserve as much meniscus as possible. Numerous studies have demonstrated a correlation between the amount of meniscus removed and the future onset of osteoarthritis.

However, in some cases, especially in the presence of complex and/or chronic lesions, meniscectomy remains the only viable surgical option. Over time, months or years later, a subgroup of patients may develop symptoms such as pain, joint swelling, and mechanical overload of the compartment that underwent meniscectomy, a condition known as post-meniscectomy syndrome..A portion of these patients will later develop knee osteoarthritis and require invasive procedures such as partial or total knee replacement.

In an attempt to treat this condition, scaffolds-collagen implants-have been developed and are arthroscopically implanted in the knee with the aim of functionally replacing the tissue removed during surgery. The goal is to reduce the incidence of long-term osteoarthritis and, consequently, the need for more invasive procedures. To date, no study has definitively demonstrated the real efficacy of these scaffolds (CMI), particularly regarding chondroprotection and the long-term onset of osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years at the time of surgery
* Both male and female patients
* Patients who underwent meniscectomy and/or CMI implantation from January 1, 1998 to December 31, 2010 at the Rizzoli Orthopedic Institute.

Exclusion Criteria:

* Patients who are no longer reachable;
* Patients who do not consent to be included in the study;
* Presence of infection or hematological, rheumatic, or hemostatic disorders at the time of evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, upon signing the informed consent, will be clinically evaluated during the follow-up visit by specialized medical personnel. A clinical examination will be performed, including the administration of subjective assessment questionnaires, and weight-bearing radiographs of the lower limbs will be conducted.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-29 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC): | 10 years after surgery
  The IKDC form is a subjective knee evaluation module that reflects the limitations on activities the individual can perform in daily life and sports, as well as the presence or absence of symptoms.
  There are three main domains in the IKDC evaluation form: Symptoms, which include pain, stiffness, swelling, and a sensation of locking; Sports and daily activities; Current knee function and function prior to injury. The questionnaire consists of 10 questions: seven items investigate the patient's symptoms, one item is focused on sports participation, one item-composed of 9 points-addresses the difficulties the patient experiences in performing daily life activities, and the last item measures the current functionality of the knee.
  The score ranges from 0 to 100, with 100 representing the absence of limitations and symptoms, indicating an excellent outcome; the further away from this score, the worse the result, which can be divided into four groups

SECONDARY OUTCOMES:
Lysholm Knee Score | 10 years after surgery
  It is a validated measurement scale that assesses knee functionality through 8 items, allowing the evaluation of the knee's condition in response to the functional demands of daily activities. This assessment form is used to evaluate surgical outcomes in patients who have undergone surgery for ligament or meniscal injuries of the knee. The final score is obtained by summing the various scores from different items, ranging from 0 to 100.
  The scores are divided into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64).
VAS | 10 years after surgery
  It is a unidimensional, quantitative numeric pain rating scale with 10 points; the scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that precise moment. 0 means no pain, and 10 indicates the worst possible pain
SF-36 (Short Form-36 Health Survey) | 10 years after surgery
  It is the most well-known and widely used health-related quality of life measurement tool in international literature. It assesses different health concepts through 36 multiple-choice questions, with the data aggregated into 8 scales that evaluate: physical activity, role and physical health, physical pain, general health, vitality, social activities, role and emotional state, mental health. Additionally, there is one question regarding changes in health status over the past year.
Tegner Score | 10 years after surgery
  It allows for estimating a person's level of physical activity with a score ranging from 0 to 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as national or international level football.' This score is the most commonly used to define the level of physical activity in patients with knee disorders. In the study, the Tegner Score will be completed directly by the investigator through an interview with the patient
Radiographic evaluation | 10 years after surgery
  Clinical and imaging materials in the patient's possession will be collected to assess the potential development of osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Rizzoli Orthopedic Institute, Bologna, Bologna, Italy